CLINICAL TRIAL: NCT02725944
Title: Prediction and Detection of Occult Atrial Fibrillation in Patients After Acute Cryptogenic Stroke and Transient Ischemic Attack
Brief Title: Prediction and Detection of Occult Atrial Fibrillation in Patients After Acute Cryptogenic Stroke and TIA
Acronym: PROACTIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Loreta Skrebelyte-Strøm, MD, MD, University Hospital, Akershus
Other Study IDs: 2014/1260 D (REK)
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Cerebrovascular Stroke; Atrial Fibrillation
Keywords: Cryptogenic stroke; Occult paroxysmal atrial fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cryptogenic stroke and TIA: Implantation of ICRM in all participants.
  Interventions: Device: Implantation of ICRM

INTERVENTIONS:
Device: Implantation of ICRM — All patients will be implanted with ICRM in order to detect an occult PAF.

SUMMARY:
PROACTIA is a prospective, event-driven observational study. It aims to propose a composite scoring system in order to evaluate the risk of paroxysmal atrial fibrillation (PAF) in patients after acute cryptogenic stroke and transient ischemic attack (TIA).

DETAILED DESCRIPTION:
It will be enrolled 250 participants of both sexes within two weeks after diagnosed cryptogenic stroke and/or TIA at Akershus University Hospital, Oslo area, Norway.

Evaluation of participants' comorbidity with CHADS2-VASc score, ECG, Holter ECG, echocardiography, detection of biochemical cardiac markers and screening for obstructive sleep apnea syndrome will be performed. All participants will be monitored with a continuous cardiac rhythm during one year by implantation of implantable cardiac rhythm monitors (ICRM). All patients without high bleeding risk will get prescribed oral anticoagulants (OAC) after detection of PAF.

A biobank will be established in order to store the sampled biological material.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with cryptogenic stroke and/or TIA, in accordance to the TOAST (Trial of Org 10172 in Acute Stroke Treatment) classification.

Exclusion Criteria:

* Patients with known or newly detected AF on initial examination including 24 h Holter ECG.
* Patients on oral anticoagulants (OAC) for non-AF indications.
* Patients with strong contraindications for OAC, even if the presence of underlying AF is detected.
* Patients with atrial- or ventricular thrombi, or atheromas of the aortic arch greater than 4 mm, detected by transesophageal echocardiography.
* Patients unable to sign the informed consent or with a life expectancy due to comorbidities of less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 participants of both sexes included at Akershus University Hospital, Norway, within two weeks after diagnosed with cryptogenic stroke and/or TIA.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Detection of paroxysmal atrial fibrillation | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Loreta Skrebelyte-Strøm, Oslo, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Skrebelyte-Strom L, Saberniak J, Bjorkan Orstad E, Mykland Hilde JE, Ronning OM, Steine K. Left atrial appendage function by strain and structure is associated with thromboembolic risk in patients with cryptogenic stroke and TIA. Open Heart. 2025 May 27;12(1):e003287. doi: 10.1136/openhrt-2025-003287. PMID 40436433
- [Derived] Skrebelyte-Strom L, Ronning OM, Dahl FA, Steine K, Kjekshus H. Prediction of occult atrial fibrillation in patients after cryptogenic stroke and transient ischaemic attack: PROACTIA. Europace. 2022 Dec 9;24(12):1881-1888. doi: 10.1093/europace/euac092. PMID 35819199